CLINICAL TRIAL: NCT06193876
Title: The Effect of Petitgrain and Ylang-ylang Oil Applied Before Clinical Practice on Stress, Anxiety and Depression in Midwifery Students.
Brief Title: The Effect of Aromatherapy Before Clinical Practice on Stress, Anxiety and Depression in Midwifery Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuba Kızılkaya (Other)
Responsible Party: Sponsor-Investigator, Tuba Kızılkaya, Asst. Prof. Dr, Balikesir University
Organization: Balikesir University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20072023
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Aromatherapy; Stress; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Petitgrain group (Active Comparator): In this group petitgrain oil will be used
  Interventions: Other: Petitgrain and ylang-ylang essential oil
- Ylang-ylang group (Active Comparator): In this group ylang-ylang oil will be used
  Interventions: Other: Petitgrain and ylang-ylang essential oil
- Placebo group (Placebo Comparator): In this group water will be used
  Interventions: Other: Petitgrain and ylang-ylang essential oil

INTERVENTIONS:
Other: Petitgrain and ylang-ylang essential oil — Petitgrain and ylan-ylang essential oil will be dropped to the handchief and students will smell it 3 times in a day.

SUMMARY:
This study was planned as a randomized controlled study to determine the effects of petitgrain and ylang ylang oil applied before clinical practice on stress, anxiety and depression in midwifery students.

ELIGIBILITY:
Inclusion Criteria:

* Being a midwifery student

Exclusion Criteria:

* Having an asthma or any other respiration disease
* Trouble of smelling
* Allergies to petitgrain or ylang-ylang essential oil

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
depression level | 1 day
stress level | 1 day
anxiety level | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Osmaniye Korkut Ata University Hospital, Osmaniye, Turkey (Türkiye)